CLINICAL TRIAL: NCT05511285
Title: Improving Sleep and Learning in Rehabilitation After Stroke, Part 2
Acronym: INSPIRES-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Big Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID 16015
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Sleep; Rehabilitation; Digital; Cognitive Behavioural Therapy for Insomnia; Motor consolidation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial with two parallel study arms: (1) digital cognitive behavioural therapy for insomnia (experimental condition), and (2) treatment as usual (control condition). Randomisation will be using a 2:1 ratio (experimental:control), within minimisation of between group differences in age, sex, baseline Sleep Condition Indicator score and time since stroke.
Who Masked: Outcomes Assessor
Masking Description: Randomisation and facilitation of the intervention will be performed by a research assistant, and the person analysing the data will be blinded to group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioural: Digital cognitive behavioural therapy for insomnia (Experimental): 6-10 weeks of digital cognitive behavioural therapy for insomnia (Sleepio) delivered online.
  Interventions: Behavioral: Digital Cognitive Behavioural Therapy for Insomnia
- Treatment as usual (No Intervention): Participants will receive treatment as usual.

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioural Therapy for Insomnia — 6-10 weeks of digital cognitive behavioural therapy for insomnia (Sleepio) delivered online, in addition to usual care.
  Other Names: Sleepio
  Arms: Behavioural: Digital cognitive behavioural therapy for insomnia

SUMMARY:
This study will explore whether sleep in stroke survivors is improved with digital cognitive behavioural therapy for insomnia (Sleepio), in comparison to treatment as usual, and will explore whether changes in sleep relate to changes in overnight consolidation of motor learning.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of adult disability. Rehabilitation of movement after stroke depends on motor learning. Motor learning involves not only improvement during practice but also offline improvement, or consolidation, that occurs after practice. Consolidation of learning depends on good sleep quality. However, sleep is disrupted long-term after stroke and patients with poorer sleep show worse rehabilitation outcomes.

Cognitive behavioural therapy for insomnia (CBT) is the recommended first line treatment for sleep problems. "Sleepio" is a digital CBT programme which is effective across a range of clinical populations. This study aims to test the efficacy of digital CBT for reducing insomnia symptoms after stroke, in comparison with usual care alone. To explore the possibility that sleep interventions might enhance rehabilitation outcomes via their impact on consolidation of motor learning, the study will additionally test for differences in consolidation between groups, and explore whether changes in sleep measures are associated with changes in consolidation.

Participants will be randomised to either receive digital CBT for insomnia (in addition to usual care) or receive treatment as usual alone (2:1 treatment to control ratio). The primary outcome is the score on the 8-item Sleep Condition Indicator, 10 weeks following randomisation. Secondary outcomes include behavioural measures of overnight motor consolidation assessed as the change in motor task performance from training to retest, sleep disruption assessed with actigraphy, and depression and fatigue using the Patient Health Questionnaire (PHQ9) and the Fatigue Severity Scale respectively.

In addition to this, to explore the feasibility of delivering rehabilitation following the sleep improvement programme, an optional 4 weeks of upper limb motor training at home will be offered to all participants (regardless of group allocation) after follow-up. Outcomes of adherence to the training and upper limb function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Aged 18 years or above.
* Clinical diagnosis of stroke affecting the upper limb, with sufficient movement to perform the motor learning task
* Discharged from inpatient care
* Interest in accessing a programme with the aim of improving sleep quality
* Reliable access to the internet

Exclusion Criteria:

* Other neurological condition affecting movement (e.g. Parkinson's Disease, Multiple Sclerosis)
* Diagnosed, untreated, sleep disorder (e.g. Sleep Apnea)
* Uncontrolled seizures
* Planned inpatient admission (e.g. for rehabilitation) in the next 4 months that would impact ability to engage with the Sleepio programme
* Engagement in psychological therapy for insomnia in the past 12 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sleep Condition Indicator | 10 weeks after randomisation
  Questionnaire assessing self-reported insomnia symptoms, range 0-32, higher numbers indicate less symptoms of insomnia

SECONDARY OUTCOMES:
Change in motor performance from training to retest | 10 weeks after randomisation
  Behavioural motor consolidation assessment, assessed as accuracy (range 0-50, higher numbers indicate better accuracy of motor performance)
Patient Health Questionnaire | 10 weeks after randomisation
  Questionnaire assessing symptoms of depression, range 0-20, higher values indicate more depressive symptoms
Fatigue Severity Scale | 10 weeks after randomisation
  Questionnaire assessing fatigue, range 9-63, higher score indicates more severe fatigue
Actigraphy | 10 weeks after randomisation
  Wearable activity monitor used for assessing sleep disruption (Total Sleep Time, Wake After Sleep Onset, sleep fragmentation)

OTHER OUTCOMES:
Adherence of at home motor training | 14 weeks following randomisation
  Assessment of number of sessions performed, number of repetitions etc.
Upper limb ability | 14 weeks following randomisation
  Assessed with Action Research Arm Test, range 0-57, higher score indicates better upper limb ability
Upper limb function | 14 weeks following randomisation
  Assessed with Box and Blocks Test, scored as the number of blocks transferred in 60 seconds
Upper limb dexterity | 14 weeks following randomisation
  Assessed with Nine hole peg test, scored as the number of pegs placed in 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Melanie K Fleming, Dr, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data are available upon reasonable request
Supporting Information: Study Protocol
Time Frame: Following publication of results
Access Criteria: Available upon reasonable request

REFERENCES:
- [Derived] Weightman M, Robinson B, Fallows R, Henry AL, Kyle SD, Garratt E, Pick A, Teal R, Ajina S, Demeyere N, Espie CA, Seymour B, Johansen-Berg H, Fleming MK. Improving sleep and learning in rehabilitation after stroke, part 2 (INSPIRES2): study protocol for a home-based randomised control trial of digital cognitive behavioural therapy (dCBT) for insomnia. BMJ Open. 2023 Apr 6;13(4):e071764. doi: 10.1136/bmjopen-2023-071764. PMID 37024247